CLINICAL TRIAL: NCT01931696
Title: Clinical Assessment of Acupuncture for the Treatment of Asthma: A Randomized, Multicenter, Double-blind, Parallel-group Controlled Trial
Brief Title: Clinical Assessment of Acupuncture for the Treatment of Chronic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Municipal Health Bureau (Other Government); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYSNXD-CC-ZDYJ039
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
Keywords: Efficacy; Acupuncture; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum acupuncture (Experimental): Verum acupuncture treatment once every two days + Albuterol sulfate HFA (Ventolin®™ 100 mcg Inhalation Aerosol) as needed + Prednisone Acetate Tablets(H31020675, 5 mg oral tablet) for exacerbation
  Interventions: Device: Verum acupuncture
- Sham acupuncture (Sham Comparator): Sham acupuncture treatment once every two days + Albuterol sulfate HFA (Ventolin®™ 100 mcg Inhalation Aerosol) as needed + Prednisone Acetate Tablets(H31020675, 5 mg oral tablet) for exacerbation
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Verum acupuncture — 100 patients receive verum acupuncture treatment once every other day,choosing Dazhui(GV14), Fengmen(BL12), Feishu(BL13), needles retention for 30 minutes and no moxibustion or electrical stimulation. Patients receive verum acupuncture once every other day with a total of 20 sessions in 6 weeks. The needle brand is Hwato®™ Sterile Acupuncture Needles for Single Use.
  Arms: Verum acupuncture
Device: Sham acupuncture — 100 patients receive sham acupuncture treatment once every other day, choosing Jinsuo(DU08), Ganshu(BL18), Danshu(BL19), needles retention for 30 minutes and no moxibustion or electrical stimulation. Patients receive sham acupuncture once every other day with a total of 20 sessions in 6 weeks. The needle brand is Hwato®™ Sterile Acupuncture Needles for Single Use.
  Arms: Sham acupuncture

SUMMARY:
The purpose of this study is to assess whether acupuncture is effective in the treatment of chronic asthma.

DETAILED DESCRIPTION:
Asthma is a common chronic disease worldwide with an estimated 300 million affected individuals. In analyses of economic burden of asthma, apart from direct medical costs including hospital admissions and cost of medications, indirect, non-medical costs such as time lost from work account for a considerable part. For all but the most severe patients, the ultimate goal is to prevent symptoms, minimize morbidity from acute episodes, and prevent functional and psychological morbidity to provide a near healthy lifestyle. Although the symptoms can be controlled by drug treatment in most patients, effective low-risk, non-drug approaches such as acupuncture could constitute a significant advance in asthma management. The purpose of this study is to assess whether acupuncture is effective in the treatment of chronic asthma.

There is a 1-week screening period(-1 week) during which participants will be monitored while they use an albuterol inhaler as needed. Study visits will occur at weeks 0(Baseline), weeks 3, weeks 6. Participants will undergo a physical examination, lung function, blood and urine collection. At the Weeks 0 study visit, participants will be randomly assigned to one of the following two groups for 6 weeks of treatment:

* Group 1 will receive verum acupuncture treatment once every two days plus albuterol as needed, prednisone for exacerbation
* Group 2 will receive sham acupuncture treatment once every two days plus albuterol as needed, prednisone for exacerbation

Study visits will occur at Weeks 0, 3, 6. A physical examination, blood collection, and lung function will occur at selected visits. Questionnaires to assess asthma control and quality of life will also be completed. Throughout the study, participants will record asthma symptoms and medication usage in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild-to-moderate persistent asthma
* Forced expiratory volume in one second (FEV1) reversibility of greater than or equal to 12% following bronchodilator administration (2 puffs)
* Patients who have given written informed consent

Exclusion Criteria:

* Participation in another clinical trial 1 month prior to study entry
* Use of systemic corticosteroids 2 weeks prior to study entry
* Patients with general infection, lower respiratory infection, pulmonary tuberculosis and fungal infection 1 month prior to study entry
* Hospitalization due to acute exacerbation 3 months prior to study entry
* Patients cannot stop using forbidden drugs which include inhaled corticosteroid, theophylline, long-term β2 agonist, sodium cromoglicate, leukotrienes antagonist and anticholinergic drug
* Patients who are allergic to albuterol and corticosteroid
* Patients with severe primary diseases such as cancer, cardiovascular system, liver, kidney and hematopoietic system diseases
* Wheeze caused by pulmonary tuberculosis, bronchiectasia and cardiac insufficiency
* Patients with hyperthyroidism
* Patients with mental illness, acrasia
* Female patients in pregnancy, lactation period and planning to get pregnant during the trial
* Any significant disorder that in the investigator's opinion, might put the patients at risk or influence the study outcomes
* Acupuncture contraindications: serious allergic or infectious dermatitis and hemorrhagic diseases such as thrombocytopenic purpura and hemophilia

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Total score Change from Baseline of Asthma Control Test | Measured during the 6 week treatment period

SECONDARY OUTCOMES:
Percentage of symptom-free days | Measured during the 6 week treatment period
Usage of salbutamol and prednisone | Measured during the 6 week treatment period
Lung function(FEV1, PVC, FEV1/FVC%, FEV1/predicted%)，morning/evening PEF | Measured during the 6 week treatment period
Asthma symptom scores | Measured during the 6 week treatment period
Asthma quality of Life Questionnaire(AQLQ) | Measured during the 6 week treatment period
Total number of exacerbations that require systemic corticosteroid therapy | Measured during the 6 week treatment period
Eosinophil (EOS) count in peripheral blood, T cell classification, serum cytokine levels | Measured during the 6 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Qing Yang, Ph.D, Study Chair — Shanghai University of TCM
Locations (12):
- China (12):
  - University Hospital of Gansu Traditional Chinese Medicine, Lanzhou, Gansu
  - Kaifeng Traditional Chinese Medicine hospital, Kaifeng, Henan
  - No.3 hospital of Henan college of Traditional Chinese Medicine, Zhengzhou, Henan
  - Zhengzhou Traditional Chinese Medicine hospital, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai research institute of acupuncture and meridian，Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - Shanghai Dachang hospital, Shanghai, Shanghai Municipality
  - Longhua Hospital, Shanghai, Shanghai Municipality
  - Shanghai TCM Integrated hospital, Shanghai, Shanghai Municipality
  - Shuguang Hospital, Shanghai, Shanghai Municipality
  - Wenzhou Hospital of Traditional Chinese Medicine, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Yin LM, Wang Y, Fan L, Xu YD, Wang WQ, Liu YY, Feng JT, Hu CP, Wang PY, Zhang TF, Shao SJ, Yang YQ. Efficacy of acupuncture for chronic asthma: study protocol for a randomized controlled trial. Trials. 2015 Sep 23;16:424. doi: 10.1186/s13063-015-0947-z. PMID 26399399